CLINICAL TRIAL: NCT04277247
Title: Botulinum Toxin A (Onabotulinumtoxin A) for Foot Dystonia-associated Pain in Parkinson's Disease: A Randomized, Double-blind Placebo Control Study
Brief Title: Botulinum Toxin Type A for Foot Dystonia-associated Pain in Parkinson's Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Veronica Bruno, Clinical Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB19-1645
Record Dates: First submitted 2020-02-10; First posted 2020-02-20 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Dystonia Disorder; Parkinson Disease
MeSH Terms: conditions — Dystonic Disorders; Parkinson Disease | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: We will perform a double-blind, randomized, parallel group study evaluating the safety and efficacy of BTXA injections vs. placebo injections, targeted at painful muscles, followed by an open-label phase when all participants will receive BTXA. Subjects, caregivers, and the investigators will be blinded to assignment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Upon entry to the study, all subjects will be assigned to a subject number. Eligible subjects will be randomized to receive either BTXA injections or placebo on VISIT 1 in a double-blind manner according to a randomization schedule using computerized randomization tables as prepared by a blinded clinical nurse. All patients will receive BTXA injections on VISIT 4 in an open-label phase. The specific type of randomization used will be block randomization to ensure equal sample sizes of the BTXA and placebo groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum Toxin Type A Treatment (Experimental): Injections
  Interventions: Drug: Botulinum toxin type A
- Placebo (Placebo Comparator): Injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum toxin type A — A standardized dose will be injected in each muscle: 25 Units of BTXA in the extensor hallucis longus in 1 site, 50 Units of BTXA in the flexor digitorum brevis in 2 sites and 25 Units of BTXA in the tibialis posterior in 1 site.
  Other Names: BTXA
  Arms: Botulinum Toxin Type A Treatment
Drug: Placebo — 0.9% saline placebo injection
  Other Names: Saline
  Arms: Placebo

SUMMARY:
To study the effects of Botulinum toxin type A (BTXA) in the treatment of foot dystonia-associated pain in Parkinson's disease

DETAILED DESCRIPTION:
Dystonia-associated pain, particularly in the lower limbs is the second most common type of pain in Parkinson's disease (PD). Involuntary muscle contractions that cause slow repetitive movements or abnormal postures are common. The movements may be painful and present in different ways, from just foot inversion or hallux extension to complex forms. They may affect the quality of life of patients in different ways during both ON and OFF periods. Cures for foot dystonia symptoms in PD are not yet available. Yet, improving pain symptoms can improve patients' quality of life. BTXA has been proposed as a safe and useful option for the treatment of PD patients affected by foot dystonia as it could improve symptoms locally without modifying any antiparkinsonian medications. Injected into muscles, BTXA could reduce rigidity, stiffness and improve abnormal postures that may cause foot pain. Recognizing different uses of BTXA will help to understand the symptomatic treatment for each patient in any stage of the disease. The results will help doctors to use new tools to treat foot-dystonia pain in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with PD according to the MDS Clinical diagnostic criteria for Parkinson's disease
* Participants with foot dystonia not responding to antiparkinsonian agents or changes in antiparkinsonian medications schedule sufficiently as per Movement Disorders Specialist. Subjects with bilateral foot dystonia will be injected in the side where the symptoms are more severe.
* BTXA treatment naïve subjects or not received any within the last six months (including other indications).
* Stable PD and pain medications for at least 30 days.
* Competence to self-report pain severity in the King's Parkinson's disease pain scale (KPPS) and a Likert Visual Analogue Scale (VAS)

Exclusion Criteria:

* Subjects with a primary cause of pain in the lower limbs unrelated to PD foot dystonia and associated with another medical condition, e.g. severe arthritis.
* Subjects that because of the severity or refractory pain are under an unfixed analgesic schedule.
* Subjects who are unable to self- report pain severity in the selected scales. Patients that may require a translator or are illiterate will be included as long as they can self-report pain severity.
* Subjects who are undergoing acute infections or other acute intercurrence.
* Any contraindication to receiving BTXA injections:

  1. Subjects who are hypersensitive to any BTXA or any ingredient in the formulation or component of the container (Clostridium Botulinum toxin type A neurotoxin complex 900 kD, Human Serum Albumin and Sodium Chloride).
  2. The presence of infection at the proposed injection site(s).

We decided to exclude patients with high risk cardiovascular disease in the case of severe orthostatic hypotension occurring secondary to the BTXA injections (reported in less than 1% of treated cases). Systemic toxic effects of BTXA are rarely reported and most of the cases in the literature are children. In order to absolutely avoid this potential complication, we will exclude patients who report sickness/infections during the study visit

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in King's Parkinson's disease pain scale score | 6 and 12 weeks during the parallel group phase and at 24 weeks during the open-label phase
  The measure foot dystonia-associated pain change perceived by the patients. The scale is composed of 14 questions exploring the frequency and severity of different pain syndromes that are frequently observed in Parkinson's disease patients, which can be summed to form an overall pain intensity score. Each item is scored by severity (0-3) multiplied by frequency (0-4), resulting in a subscore of 0 to 12, with a total possible score range from 0 to 168. Higher scores are indicative of worse outcomes.
Change in Likert Visual Analogue Scale | 6 and 12 weeks during the parallel group phase and at 24 weeks during the open-label phase
  The measure of foot dystonia-associated pain change perceived by the patients. The most simple Likert Visual Analogue Scale is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best). There are no numerical values on this scale however, a positioning towards the left of the scale indicates a worse outcome.

SECONDARY OUTCOMES:
Change in Clinical Global Impression Scale | 6 and 12 weeks during the parallel group phase
  Changes in scores on the Clinical Global Impression (CGI) scale. CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients).CGI scores range from 1 (very much improved) through to 7 (very much worse). Treatment response ratings should take account of both therapeutic efficacy and treatment-related adverse events and range from 0 (marked improvement and no side-effects) and 4 (unchanged or worse and side-effects outweigh the therapeutic effects). Each component of the CGI is rated separately; the instrument does not yield a global score.
Change in Movement Disorder Society Unified Parkinson Disease Rating Scale Parts 1-4 (MDS-UPDRS) ON medication | 6 and 12 weeks during the parallel group phase
  Measures changes of symptom severity, treatment response and the efficacy of treatments. Part 1 (non-motor experiences of daily living), Part 2 (motor experiences of daily living), Part 3 (motor examination) and Part 4 (motor complications). The maximum score for all the parts is 272. Higher scores are indicative of worse outcomes.
Change in gait | 6 and 12 weeks during the parallel group phase
  Changes in gait will be assessed according to the sections Postural Instability/Gait Difficulty sub-score of the Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS UPDRS) part 3. Higher score indicative or worse outcomes.
Change in Parkinson's Disease 39 item Quality of life questionnaire | 6 and 12 weeks during the parallel group phase
  This 39 - item questionnaire assesses Parkinson's disease-specific health-related quality over the last month. It assesses how often patients experience difficulties across 8 quality of life dimensions including functioning and well being. Scores can range from 0 to 100. The higher score is indicative of worse quality of life.
Number of adverse events | 6 and 12 weeks during the parallel group phase. Adverse events will be also documented 24 weeks during the open-label phase.
  Adverse events assessed for safety purposes at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Bruno, MD, MPH, Principal Investigator — University of Calgary
Locations (1):
- Movement Disorder Program, Foothills Medical Center, Alberta Health Services, Calgary, Alberta, Canada